CLINICAL TRIAL: NCT01219673
Title: A Study of Reducing the Symptom Burden Produced by Chemoradiation Treatment for Head and Neck Cancer
Brief Title: Symptom Burden in Head and Neck Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Low accrual.
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2009-0517; R01 026582-26 (Other Grant/Funding Number: NCI)
Record Dates: First submitted 2010-10-11; First posted 2010-10-13 (Estimated); Results first posted 2015-02-10 (Estimated); Last update posted 2015-02-10 (Estimated); Status verified 2015-01

CONDITIONS: Head And Neck Cancer
Keywords: Epithelial carcinoma; Oropharynx; Larynx; Symptom-management; Chemoradiation; Placebo; Armodafinil; Nuvigil; Bupropion; Wellbutrin; Wellbutrin SR; Zyban; Minocycline; Dynacin; Minocin; Minocin PAC; Myrac; Solodyn
MeSH Terms: conditions — Head and Neck Neoplasms; Carcinoma; Laryngeal Diseases; cyclopia sequence | interventions — Modafinil; Minocycline; Bupropion

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- Placebo (Placebo Comparator): Placebo by mouth 2 times every day.
  Interventions: Other: Placebo
- Armodafinil (Experimental): Armodafinil 150 mg by mouth once a day.
  Interventions: Drug: Armodafinil
- Minocycline (Experimental): Minocycline 100 mg by muth two times a day.
  Interventions: Drug: Minocycline
- Bupropion (Experimental): Bupropion 100 mg by mouth two times a day.
  Interventions: Drug: Bupropion
- Armodafinil + Minocycline (Experimental): Armodafinil 150 mg by mouth once a day.
  Minocycline 100 mg by mouth two times a day.
  Interventions: Drug: Armodafinil; Drug: Minocycline
- Armodafinil + Bupropion (Experimental): Armodafinil 150 mg by mouth once a day.
  Bupropion 100 mg by mouth two times a day.
  Interventions: Drug: Armodafinil; Drug: Bupropion
- Minocycline + Bupropion (Experimental): Minocycline 100 mg by muth two times a day.
  Bupropion 100 mg by mouth two times a day.
  Interventions: Drug: Minocycline; Drug: Bupropion
- Armodafinil + Minocycline + Bupropion (Experimental): Armodafinil 150 mg by mouth once a day.
  Minocycline 100 mg by muth two times a day.
  Bupropion 100 mg by mouth two times a day.
  Interventions: Drug: Armodafinil; Drug: Minocycline; Drug: Bupropion

INTERVENTIONS:
Other: Placebo — 1 by mouth twice a day.
  Arms: Placebo
Drug: Armodafinil — 150 mg by mouth once a day.
  Other Names: Nuvigil
  Arms: Armodafinil; Armodafinil + Bupropion; Armodafinil + Minocycline; Armodafinil + Minocycline + Bupropion
Drug: Minocycline — 100 mg by mouth twice a day.
  Other Names: Dynacin; Minocin; Minocin PAC; Myrac; Solodyn
  Arms: Armodafinil + Minocycline; Armodafinil + Minocycline + Bupropion; Minocycline; Minocycline + Bupropion
Drug: Bupropion — 100 mg by mouth twice a day.
  Other Names: Wellbutrin; Wellbutrin SR; Zyban
  Arms: Armodafinil + Bupropion; Armodafinil + Minocycline + Bupropion; Bupropion; Minocycline + Bupropion

SUMMARY:
The goal of this clinical research study is to compare armodafinil, bupropion, and minocycline when given alone or in combination. Researchers want to learn about the safety and level of effectiveness of these drugs in controlling symptoms, such as the side effects of chemoradiation, when given to patients with head and neck cancer.

DETAILED DESCRIPTION:
The Study Drugs:

It is not known which study drug or combination of study drugs is better at reducing side effects patients may experience during chemoradiation therapy. For this reason, researchers have chosen 3 study drugs that may help to reduce side effects such as fatigue, pain, sleep disturbance, difficulty swallowing, and lack of appetite. The study drugs will be tested alone and in combination with each other.

* Armodafinil is designed to prevent excessive sleepiness.
* Bupropion and minocycline each may reduce inflammation, which may help to reduce other symptoms. Bupropion is a drug for depression. Minocycline is an antibiotic (a drug to treat infection).

Study Groups:

If you agree to take part in this study, you will be randomly assigned (as in the roll of dice) to 1 of 8 groups. You may be assigned to receive no study drugs, 1 study drug, a combination of 2, or all 3 of the study drugs.

During this study, you may receive 1 or more placebos. A placebo looks like the study drug(s) but has no active ingredients. There is a chance that you will be in a group that does not receive any study drugs at all. The study drugs are being tested to learn if they can help control symptoms. All participants will be able to receive standard care for head and neck cancer outside of the study.

Neither you nor the study staff will know if you are receiving the study drugs and/or the placebo(s). However, if needed for your safety, the study staff will be able to find out which study drug(s) you are receiving.

Study Drug Administration:

You will take the study drugs/placebos 2 times every day for up to 10 weeks. You will take 1 or more study drug(s) or placebos by mouth each time, as instructed by the study doctor. If you have trouble swallowing the study drugs/placebos, they can be crushed just before taking them. You will be given information sheets on how to take the study drugs/placebos.

You will be given a daily diary to write down when you take the study drugs/placebos. You should bring your study drugs/placebos to the clinic to every study visit. You should also bring your diary to every study visit.

Symptom Questionnaire:

Throughout the study, you will be asked to fill out a symptom questionnaire. You will be asked about symptoms you may be experiencing and how they may be interfering with your daily activities. When you are in the clinic, the questionnaire can be completed by paper and pen with the study staff or by entering your answers into a computer. When you are away from the clinic, the questionnaire may be completed either through a phone call with the study staff or through a phone call from the interactive voice response (IVR) system. The symptom questionnaire will take up to 5 minutes each time. The study staff will give you the information you need to complete the questionnaire through the IVR system.

During Weeks 1-10, you will complete the symptom questionnaire 2 times a week. During Weeks 11-16, you will complete the symptom questionnaire 1 time a week.

If you would like, you can fill out a paper version of the questionnaire instead of using the phone system.

Study Visits:

Before you begin chemoradiation:

* You will fill out 6 questionnaires about pain and other symptoms, your mood, your tobacco and alcohol use, and the quality of your life. This should take about 15 minutes.
* You will have a blood coagulation test, called PT-INR, to make sure your blood clots normally.
* If you are a woman who is able to become pregnant, you will have a urine pregnancy test. The study staff will give you the pregnancy test kit at your scheduled visit, and will review and record the results of the test before your study prescriptions are filled by the pharmacy. This will also be done at about Weeks 4 and 7, at the first follow-up visit after radiation treatment, and 30 days after the study drugs are stopped.

At about Week 4 of chemoradiation:

* You will fill out 1 quality-of-life questionnaire. This should take about 2-3 minutes.
* You will be asked three questions about smoking after the start of chemoradiation therapy.
* You will have a blood coagulation test, called PT-INR, to make sure your blood clots normally.

During the last week of chemoradiation (about Week 7):

-You will fill out 3 questionnaires about your symptoms, mood, and quality of life. This should take about 10 minutes.

After about Week 7, the study staff will call you 2 times per week to check on you until Week 10. This phone call should last only a few minutes. If you have experienced several side effects from chemoradiation, this phone call may take longer.

At about Week 10 and at your first follow-up visit after your chemoradiation treatment:

* You will fill out 3 questionnaires about your symptoms, mood, and quality of life.
* You will fill out 2 questionnaires that ask about your smoking history and changes in your tobacco use during the study. This will take a few minutes.
* You will be asked to fill out another questionnaire that asks about your satisfaction with the study drug(s). For example, you will be asked if you thought the study drugs helped to control the symptoms, if you would recommend the study drugs to other patients, and if you had problems taking the study drugs. This will take a few minutes.
* In addition, at your first follow-up visit after your chemoradiation treatment, you will have a blood coagulation test, called PT INR, to make sure your blood clots normally.

Length of Study:

You will take the study drug(s)/placebo for up to 10 weeks, if the doctor thinks it is in your best interest. You will fill out the symptom questionnaires by phone until 16 weeks. You will no longer be able to take the study drug(s)/placebo if you experience intolerable side effects.

This is an investigational study. Armodafinil is FDA approved and commercially available for the treatment of excessive sleepiness. Bupropion is FDA approved and commercially available for the treatment of depression. Minocycline is FDA approved and commercially available for the treatment of bacterial infection. The different possible combinations of these drugs being used in this study are investigational.

Up to 32 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a pathologically proven diagnosis of epithelial carcinoma of the oropharynx, nasopharynx, hypopharynx, larynx, or oral cavity being treated at MDACC.
2. Patients >/= 18 years old and </= 65 years old.
3. Patients with the above cancers scheduled to receive definitive concurrent chemoradiation over 6 - 7 weeks.
4. Patients who speak English (due to the novel research and its complexity, we are only accruing English speaking patients to the protocol)
5. Patients must agree to discontinue any current herbal supplement use, and refrain from taking any herbal supplement while on protocol.
6. Patients must be willing and able to review, understand, and provide written consent.
7. Women of childbearing potential (women who are not postmenopausal for at least one year and are not surgically sterile) must have negative urine pregnancy test..
8. Sexually active males and females must agree to use birth control or abstinence for the duration of the trial.

Exclusion Criteria:

1. Patients who are taking medications or have conditions that potentially preclude use of any study medications or interventions as determined by the treating physician
2. Patients taking CHANTIX (smoking cessation medication)
3. Patients who are enrolled in other symptom management trial or receiving active therapy as part of a treatment clinical trial.
4. Bile duct obstruction or cholelithiasis
5. History of clinically significant cutaneous drug reaction, or a history of clinically significant hypersensitivity reaction, including multiple allergies or drug reaction
6. Pre-existing psychosis or bipolar disorder. Patients with major depressive disorder or severe depression (a score of 13 or greater on the BDI Fast Screen (BDI-FS) will be excluded. If this is the case, we will notify their treating physician for appropriate management or referral.
7. Pre-existing renal impairment: The screening cut off for serum creatinine > the upper limit of normal, will be done by the oncologist to qualify for chemoradiation.
8. Pre-existing hepatic impairment: The screening for total bilirubin > 1.5 times the upper limit of normal will be done by the oncologist to qualify for chemoradiation. The screening for >2 times the upper limit of normal hepatotoxicity: Alkaline phosphatase (ALP) and Alanine aminotransferase (ALT) will be done by the oncologist to qualify for chemoradiation.The screening results for Aspartate aminotransferase (AST) must be < 2 times the upper limit of normal if available in the medical records.
9. Pre-existing Tourette's syndrome
10. Seizure disorder
11. Anorexia/bulimia in past two months
12. Use of monoamine oxidase (MAO inhibitors) within 14 days
13. Patients undergoing abrupt discontinuation of ethanol or sedatives (including benzodiazepines)
14. Patients currently taking any of the study drugs
15. Hypersensitivity to any tetracyclines
16. Patients on anticoagulants (ie warfarin/heparin)
17. Patients with INR > 1.5.
18. Patients being treated with concurrent cetuximab chemotherapy with radiation therapy.
19. Patients currently receiving any tetracycline family antibiotic or within the previous past 14 days before chemoradiation.
20. Previous radiation therapy for a cancer in the head and neck region.
21. Patients with a history of cardiac disease, including angina and cardiac ischemia, left ventricular hypertrophy, myocardial infarction, and mitral valve prolapse.
22. Patients taking antifungals, antiretrovirals, and macrolides that are strong CYP3A4 strong inhibitors including indinavir, nelfinavir, ritonavir, clarithromycin, itraconazole, ketoconazole, and nefazodone.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2013-03; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David I. Rosenthal, MD, MA, BA, Principal Investigator — UT MD Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Vita G, Compri B, Matcham F, Barbui C, Ostuzzi G. Antidepressants for the treatment of depression in people with cancer. Cochrane Database Syst Rev. 2023 Mar 31;3(3):CD011006. doi: 10.1002/14651858.CD011006.pub4. PMID 36999619
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: March 21, 2013 to June 25, 2013. All recruitment occurred at The University of Texas (UT) MD Anderson Cancer Center.
Pre-assignment Details: Due to study design changes and restrictive eligibility criteria, study enrollment was low therefore study terminated early with only one participant enrolled.
Groups:
- Armodafinil + Minocycline: Armodafinil 150 mg by mouth once a day.
  Minocycline 100 mg by mouth two times a day.
  Armodafinil: 150 mg by mouth once a day.
  Minocycline: 100 mg by mouth twice a day.
- Armodafinil + Bupropion: Armodafinil 150 mg by mouth once a day.
  Bupropion 100 mg by mouth two times a day.
  Armodafinil: 150 mg by mouth once a day.
  Bupropion: 100 mg by mouth twice a day.
- Minocycline + Bupropion: Minocycline 100 mg by muth two times a day.
  Bupropion 100 mg by mouth two times a day.
  Minocycline: 100 mg by mouth twice a day.
  Bupropion: 100 mg by mouth twice a day.
- Armodafinil + Minocycline + Bupropion: Armodafinil 150 mg by mouth once a day.
  Minocycline 100 mg by muth two times a day.
  Bupropion 100 mg by mouth two times a day.
  Armodafinil: 150 mg by mouth once a day.
  Minocycline: 100 mg by mouth twice a day.
  Bupropion: 100 mg by mouth twice a day.
Period: Overall Study
Arm/Group | Placebo | Armodafinil | Minocycline | Bupropion | Armodafinil + Minocycline | Armodafinil + Bupropion | Minocycline + Bupropion | Armodafinil + Minocycline + Bupropion
Started | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Study halted due to low enrollment (one participant). No analysis completed.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Armodafinil | Minocycline | Bupropion | Armodafinil + Minocycline | Armodafinil + Bupropion | Minocycline + Bupropion | Armodafinil + Minocycline + Bupropion | Total
Number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Age, Categorical [Number; unit: participants]
  <=18 years |  |  | 0 |  |  |  |  |  | 0
  Between 18 and 65 years |  |  | 1 |  |  |  |  |  | 1
  >=65 years |  |  | 0 |  |  |  |  |  | 0
Gender [Number; unit: participants]
  Female |  |  | 0 |  |  |  |  |  | 0
  Male |  |  | 1 |  |  |  |  |  | 1
Region of Enrollment [Number; unit: participants]
  United States |  |  | 1 |  |  |  |  |  | 1

OUTCOME MEASURES:

1. Primary Outcome: Treatment Effects on 5 Selected Symptoms (Average MDASI-HNC Scores)
Description: Treatments ability to reduce values of 5 symptoms comprised of MD Anderson Symptom Inventory (MDASI)-Head and Neck Cancer (HNC) scores for fatigue, difficulty swallowing, sleep disturbance, pain, and lack of appetite collected during the 10 weeks of chemoradiation treatment. symptoms that are caused by their disease or by their treatment. Symptom severity score is comprised of average of the five above MDASI core items (fatigue, difficulty swallowing, sleep disturbance, pain, and lack of appetite). Participants were asked to rate severity of each symptom at their worst in last 24 hours; each item rated from 0 to 10, with 0 = symptom not present and 10 = as bad as you can imagine. Total average score range: 0 to 10. Lower scores indicated better outcome.
Time Frame: 10 weeks
Population: No analysis was completed. Study terminated with low enrollment.
Arm/Group | Placebo | Armodafinil | Minocycline | Bupropion | Armodafinil + Minocycline | Armodafinil + Bupropion | Minocycline + Bupropion | Armodafinil + Minocycline + Bupropion
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: The study was active for 9 months. Participants seen weekly during treatment; continuing toxicity and other clinical variables collected by research staff at weeks 4, 7, 10, through first follow-up visit post radiation treatment.
Arm/Group | Placebo | Armodafinil | Minocycline | Bupropion | Armodafinil + Minocycline | Armodafinil + Bupropion | Minocycline + Bupropion | Armodafinil + Minocycline + Bupropion
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/1 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/1 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Analysis was not possible due to early termination with only one participant accrued.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes